CLINICAL TRIAL: NCT05453773
Title: Waterpipe Tobacco Additives and Their Effect on Human Puffing Behavior, Toxicant Exposures, Pulmonary Function, and Appeal
Brief Title: Hookah Additive Research to Inform Product Standards
Acronym: HARPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Ohio State University (Other); National Cancer Institute (NCI) (NIH); Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Marielle Brinkman, Research Professor, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: OSU-22158; NCI-2022-05156 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R01CA255563 (NIH)
Record Dates: First submitted 2022-07-01; First posted 2022-07-12 (Actual); Results first posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Tobacco-Related Carcinoma
MeSH Terms: interventions — Smoking Devices

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Tobacco flavor preparation; High Sweetness, High Humectant (tobacco smoking) (Experimental): Participants smoke 1 of 4 waterpipe tobacco preparations over 45-60 minutes over 4 sessions, separated by at least 1 week. Questionnaires administered.
  Interventions: Other: Questionnaire Administration; Behavioral: Tobacco Smoking
- Tobacco flavor preparation; High Sweetness, Medium Humectant (tobacco smoking) (Experimental): Participants smoke 1 of 4 waterpipe tobacco preparations over 45-60 minutes over 4 sessions, separated by at least 1 week. Questionnaires administered.
  Interventions: Other: Questionnaire Administration; Behavioral: Tobacco Smoking
- Tobacco flavor preparation; Medium Sweetness, High Humectant (tobacco smoking) (Experimental): Participants smoke 1 of 4 waterpipe tobacco preparations over 45-60 minutes over 4 sessions, separated by at least 1 week. Questionnaires administered.
  Interventions: Other: Questionnaire Administration; Behavioral: Tobacco Smoking
- Tobacco flavor preparation; Medium Sweetness, Medium Humectant (tobacco smoking) (Experimental): Participants smoke 1 of 4 waterpipe tobacco preparations over 45-60 minutes over 4 sessions, separated by at least 1 week. Questionnaires administered.
  Interventions: Other: Questionnaire Administration; Behavioral: Tobacco Smoking

INTERVENTIONS:
Other: Questionnaire Administration — Ancillary studies
Behavioral: Tobacco Smoking — Smoke waterpipe tobacco
  Other Names: Smoking; Tobacco, Smoking

SUMMARY:
This clinical trial evaluates how the content of waterpipe (WP) tobacco affects the appeal, puffing behavior, and toxicity of WP tobacco smoking. The data from the proposed study will provide direct links between WP tobacco's primary additives (sugars and humectants), CO and nicotine biomarkers, smoker preferences, perceptions of harm and puffing behaviors, and the subsequent range of toxicant exposures associated with these additives and behaviors. Study outcomes include waterpipe puffing behaviors, exhaled carbon monoxide levels, nicotine uptake, spirometry, sensory perceptions, smoking appeal, and risk perception. Waterpipe tobacco smoking is often the first combustible tobacco product tried by adolescents and young adults, possibly due to the widespread availability of heavily sweetened waterpipe tobacco and the perception that waterpipe smoking is a safer alternative to cigarette smoking. However, waterpipe tobacco smoking is associated with lung disease, carbon monoxide poisoning, and precursor conditions for oral and other cancers in adolescents and young adults. There is currently little data available on how the primary additives (by weight) in waterpipe tobacco affect puffing behaviors, toxicant exposures, pulmonary function and appeal. This clinical trial uses established waterpipe tobacco smokers, four investigational tobacco products with precisely manipulated levels of humectants and natural sugars in a single-blind, crossover (repeated measures) study design to determine how waterpipe tobacco additives effect human puffing behavior, nicotine uptake, flavor perceptions, lung function, and biomarkers of exposure.

DETAILED DESCRIPTION:
Currently there are no regulations governing the content of WP tobacco. Because mandated changes in tobacco content may lead to unintended consequences that ultimately result in public health declines, human use behaviors must be well understood prior to implementing regulatory product standards. The proposed study will include preparing and characterizing the content of 4 investigational tobacco products (ITPs) (Aim 1); characterizing the mainstream smoke toxicant emissions from machine smoking the 4 ITPs using a single, established puffing regimen (Aim 2); measuring human puffing behavior, general harm and specific health risk and flavor perceptions, lung function, and biomarkers of exposure in a group of established WP smokers smoking the 4 ITPs in the laboratory (Aim 3), and estimating toxicant exposure ranges using machine smoking and puffing regimens derived from the human laboratory testing (Aim 4).

The clinical trial (Aim 3) will focus on using a group of established adult and young adult WP smokers, a cross-over study design, CO and nicotine biomarkers, spirometry, cutting edge psychophysical measurement tools, and risk perception instruments to map the relationship between sensory experiences and preferences of sweetness and flavor to specific additive content in WP tobacco that affect these experiences, preferences, acute health effects, and toxicant exposures. Study subjects will participate in a series of 4 clinic sessions, each visit separated by at least a week, in which they smoke one of 4 tobacco preparations (single-blind) using a research grade waterpipe in a randomly assigned sequence in a smoking room with sufficiently controlled ventilation rate to keep ambient air CO levels below 25 ppm. Exhaled CO, whole blood samples and spirometry measures will be collected before and immediately after the smoking session. Taste perceptions, liking/disliking, and risk perceptions will be determined via questionnaires before, during, and after smoking.

ELIGIBILITY:
Inclusion Criteria:

* Sufficient understanding of consent form and study procedures
* Age 21-50 years old
* Experienced WP smokers defined as having smoked a WP at least 3 times per month in the last month
* Willing/able to abstain from nicotine product use for at least 12 hours prior to the laboratory visits
* Willing to attend four laboratory sessions at the same time of day lasting approximately 3 hours (h) each
* Read and speak English

Exclusion Criteria:

* Evident intoxication on any visit
* Exhaled breath CO > 10 ppm
* Pregnancy (known or suspected), trying to become pregnant, breastfeeding, unwillingness to use contraception for the duration of the study
* Significant smoking-related disease (by history)
* Any of the following in the past 30 days (self-report):

  * Uncontrolled asthma or asthma that is worse than usual
  * Severe respiratory allergies, such as wheezing, coughing, shortness of breath when exposed to known allergens
  * Acute upper or lower respiratory illnesses like the flu, common cold, or pneumonia
  * Any other serious lung infection or disease, such as tuberculosis, cystic fibrosis, or lung cancer
  * Hospitalization for difficulty breathing
* Currently engaging in a WP tobacco smoking quit attempt

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2022-06-19 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marielle C Brinkman, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Population: Full population of participants participating in the randomized crossover trial. Over a series of four laboratory sessions each participant received all four treatments in a randomized order, one treatment per session.
Period: Overall Study
Arm/Group | Overall Population
Started | 54
High Humectant, High Sweetness | 47
High Humectant, Medium Sweetness | 46
Medium Humectant, High Sweetness | 46
Medium Humectant, Medium Sweetness | 48
Completed | 45
Not Completed | 9
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 3
Not completed — Difficult Blood Draw | 3

BASELINE CHARACTERISTICS:
Population: 3 participants were unable to complete any study visits due to difficult blood draws; these participants are excluded here
Groups:
- Overall Population: Population of randomized participants who fully completed at least one study visit
Arm/Group | Overall Population
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.55 (4.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 19
  White | 18
  More than one race | 2
  Unknown or Not Reported | 5
Age when first tried Waterpipe [Mean (Standard Deviation); unit: years] | 18.69 (4.47)

OUTCOME MEASURES:

1. Primary Outcome: Change in Exhaled Breath Carbon Monoxide (CO)
Description: Change from baseline exhaled breath carbon monoxide (boost). CO was collected before and immediately after each smoking session with a handheld electrochemical cell.
Time Frame: Approximately 30 to 90 minutes
Measure: Mean (Standard Deviation); unit: ppm
Groups:
- High Humectant, High Sweetness: Tobacco Preparation: High Humectant, High Sweetness
- High Humectant, Medium Sweetness: Tobacco Preparation: High Humectant, Medium Sweetness
- Medium Humectant, High Sweetness: Tobacco Preparation: Medium Humectant, High Sweetness
- Medium Humectant, Medium Sweetness: Tobacco Preparation: Medium Humectant, Medium Sweetness
Arm/Group | High Humectant, High Sweetness | High Humectant, Medium Sweetness | Medium Humectant, High Sweetness | Medium Humectant, Medium Sweetness
Number analyzed (Participants) | 47 | 46 | 46 | 48
ppm | 80.1 (76.9) | 40.8 (28.5) | 62.5 (49.5) | 45.5 (31.1)

2. Primary Outcome: Change in Plasma Nicotine
Description: Change from baseline plasma nicotine (boost): Whole blood was collected before and immediately after each smoking session, separated, and plasma layer transferred and stored at -80 °C until analysis for nicotine according to validated methods using LC-MS/MS.
Time Frame: Approximately 30 to 90 minutes
Population: Participants who attended their study visit and were able to provide a plasma sample
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | High Humectant, High Sweetness | High Humectant, Medium Sweetness | Medium Humectant, High Sweetness | Medium Humectant, Medium Sweetness
Number analyzed (Participants) | 45 | 43 | 44 | 44
ng/mL | 5.1 (3.7) | 8.3 (8.4) | 6.9 (6.2) | 8.8 (8.7)

3. Primary Outcome: Change in Forced Vital Capacity (FVC)
Description: Spirometer measurements will be collected - change in forced vital capacity (FVC) (post-pre).
Time Frame: Approximately 30 to 90 minutes
Population: Spirometry was not collected at the end of the session for 1 participant during their medium humectant, high sweetness study visit.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | High Humectant, High Sweetness | High Humectant, Medium Sweetness | Medium Humectant, High Sweetness | Medium Humectant, Medium Sweetness
Number analyzed (Participants) | 47 | 46 | 45 | 48
Liters | -0.11 (0.44) | -0.03 (0.26) | 0.02 (0.16) | 0.05 (0.33)

4. Primary Outcome: Change in Forced Expiratory Volume in 1 Second (FEV1)
Description: Spirometer measurements will be collected - change in forced expiratory volume in 1 second (FEV1) (post-pre)
Time Frame: Approximately 30 to 90 minutes
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | High Humectant, High Sweetness | High Humectant, Medium Sweetness | Medium Humectant, High Sweetness | Medium Humectant, Medium Sweetness
Number analyzed (Participants) | 47 | 46 | 45 | 48
Liters | -0.05 (0.37) | -0.06 (0.22) | -0.02 (0.29) | -0.002 (0.33)

5. Primary Outcome: Change in FEV1/FVC; The Ratio of the Forced Expiratory Volume in the First One Second to the Forced Vital Capacity of the Lungs.
Description: Spirometer measurements will be collected - change in FEV1/FVC, the ratio of the forced expiratory volume in the first one second to the forced vital capacity of the lungs (post-pre).
Time Frame: Approximately 30 to 90 minutes
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | High Humectant, High Sweetness | High Humectant, Medium Sweetness | Medium Humectant, High Sweetness | Medium Humectant, Medium Sweetness
Number analyzed (Participants) | 47 | 46 | 45 | 48
ratio | 0.01 (0.05) | -0.01 (0.04) | -0.01 (0.06) | -0.01 (0.08)

6. Primary Outcome: Change in Peak Expiratory Flow (PEF)
Description: Spirometer measurements will be collected - change in peak expiratory flow (PEF) (post-pre).
Time Frame: Approximately 30 to 90 minutes
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Liters / second
Arm/Group | High Humectant, High Sweetness | High Humectant, Medium Sweetness | Medium Humectant, High Sweetness | Medium Humectant, Medium Sweetness
Number analyzed (Participants) | 47 | 46 | 45 | 48
Liters / second | -0.33 (1.12) | -0.38 (1.05) | -0.41 (1.03) | -0.33 (1.27)

7. Primary Outcome: Change in Forced Expiratory Flow at 25-75% of FVC
Description: Spirometer measurements will be collected - change in forced expiratory flow at 25-75% of FVC (post-pre).
Time Frame: Approximately 30 to 90 minutes
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: L/s
Arm/Group | High Humectant, High Sweetness | High Humectant, Medium Sweetness | Medium Humectant, High Sweetness | Medium Humectant, Medium Sweetness
Number analyzed (Participants) | 47 | 46 | 45 | 48
L/s | 0.05 (0.14) | -0.03 (0.14) | 0.0001 (0.16) | -0.01 (0.23)

8. Primary Outcome: Tobacco Use History
Description: Ever use of tobacco products, assessed at the first study visit
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Population
Number analyzed (Participants) | 51
Participants
  Cigarettes | 30
  Cigars | 36
  Cigarillos or Little Cigars | 30
  Smokeless Tobacco | 13
  Juul or Other Brands of Pod-like Electronic Cigarettes | 31
  Non-Juul Electronic Cigarettes | 29
  Pipe Tobacco | 19
  Bidis or Kreteks | 1

9. Primary Outcome: Nicotine Dependence (HONC)
Description: Hooked on Nicotine Checklist (HONC) comprised of 10 "Yes" or "No" questions, assessed on the first study visit. Scores range from 0 to 10 with higher scores indicating greater nicotine dependence.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Overall Population
Number analyzed (Participants) | 51
score on a scale | 2.16 (2.61)

10. Primary Outcome: Nicotine Dependence (LWDS)
Description: Lebanese Waterpipe Dependence Scale (LWDS) comprised of twelve questions and assessed on the first study visit. LWDS values range from 0 to 36 where higher sores indicate greater nicotine dependence.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Overall Population
Number analyzed (Participants) | 51
score on a scale | 7.88 (4.28)

11. Primary Outcome: General Harm and Health Risk Perceptions
Description: Assessed using harm/health risk perceptions questionnaire. General harm is rated after the smoking session on a scale from 0 (no harm) to 10 (extreme harm) with higher scores indicating a greater perceived harm/health risk.
Time Frame: Post Smoking Session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Humectant, High Sweetness | High Humectant, Medium Sweetness | Medium Humectant, High Sweetness | Medium Humectant, Medium Sweetness
Number analyzed (Participants) | 47 | 46 | 46 | 48
score on a scale | 5.89 (2.03) | 6.35 (2.16) | 6.15 (2.05) | 6.13 (2.19)

12. Primary Outcome: Subjective Effects of Smoking Tobacco
Description: Direct Effects of Tobacco scale; the scale for each effect ranges from 0 (not at all) to 100 (extremely) with higher ratings indicating a greater effect of the tobacco.
Time Frame: Post Smoking Session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Humectant, High Sweetness | High Humectant, Medium Sweetness | Medium Humectant, High Sweetness | Medium Humectant, Medium Sweetness
Number analyzed (Participants) | 47 | 46 | 46 | 48
score on a scale
  Satisfying | 34.17 (29.04) | 27.24 (26.87) | 29.15 (26.00) | 26.17 (25.88)
  Pleasant | 34.60 (29.28) | 27.07 (27.94) | 26.80 (25.49) | 25.75 (24.24)
  Taste Good | 29.17 (28.58) | 19.00 (22.53) | 22.15 (23.00) | 21.85 (25.68)
  Taste Bad | 45.60 (33.48) | 56.17 (33.68) | 50.57 (33.97) | 52.08 (35.71)
  Make you Dizzy | 10.94 (15.58) | 14.46 (24.43) | 16.76 (21.25) | 18.21 (22.36)
  Calm you Down | 30.21 (30.69) | 22.65 (27.93) | 26.63 (28.97) | 26.56 (30.23)
  Feel Confused | 3.62 (9.89) | 3.30 (11.83) | 3.15 (8.31) | 3.19 (11.23)
  Help you Concentrate | 21.43 (29.82) | 13.63 (23.26) | 13.54 (25.45) | 13.56 (23.70)
  Feel More Awake | 25.66 (31.31) | 12.67 (20.82) | 18.70 (27.63) | 17.31 (25.29)
  Reduce Hunger | 17.89 (27.80) | 13.67 (23.71) | 12.11 (21.99) | 14.98 (25.19)
  Make you Sick | 4.55 (9.59) | 7.13 (16.72) | 9.33 (16.43) | 8.60 (16.86)
  Make you Sleepy | 12.43 (21.03) | 12.76 (21.36) | 12.48 (21.13) | 6.65 (16.06)
  Like to smoke another hookah right now | 25.64 (30.30) | 13.35 (21.61) | 16.09 (25.34) | 17.00 (24.23)

13. Primary Outcome: Change in Subjective Effects of Smoking Tobacco - Direct Effects of Nicotine
Description: Change in Direct Effects of Nicotine scale from baseline (post - pre). The scale for each effect ranges from 0 (not at all) to 100 (extremely) with higher ratings indicating a greater effect of the tobacco.
Time Frame: Approximately 30 to 90 minutes
Population: Data is missing for 1 participant from the High Humectant, High Sweetness and Medium Humectant, Medium Sweetness arms as they declined to respond to the pre-smoking survey items.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Humectant, High Sweetness | High Humectant, Medium Sweetness | Medium Humectant, High Sweetness | Medium Humectant, Medium Sweetness
Number analyzed (Participants) | 46 | 46 | 46 | 47
score on a scale
  Nauseous | 0.33 (9.45) | -0.07 (11.98) | -0.02 (13.18) | 2.94 (13.02)
  Dizzy | 0.96 (9.72) | 0.89 (13.17) | 2.57 (10.24) | 2.57 (11.98)
  Lightheaded | 6.80 (13.95) | 0.74 (13.92) | 4.91 (17.73) | 4.19 (14.75)
  Nervous | -2.13 (5.96) | -2.09 (9.13) | -0.67 (3.39) | 1.23 (6.85)
  Sweaty | 0.28 (6.90) | -1.20 (8.62) | 1.09 (7.31) | 1.51 (11.37)
  Headache | -0.93 (14.04) | -1.48 (18.86) | 1.96 (13.96) | 1.21 (11.66)
  Excessive Salivation | 3.15 (11.08) | -0.67 (13.21) | 1.43 (9.95) | 2.81 (12.65)
  Heart Pounding | 0.30 (6.15) | 0.02 (9.07) | 0.20 (5.95) | 2.13 (8.83)
  Confused | -0.30 (2.14) | -0.76 (8.39) | 0.28 (3.89) | 0.23 (3.30)
  Weak | -1.20 (7.17) | 0.39 (10.36) | 1.50 (10.94) | 0.81 (6.54)

14. Primary Outcome: Change in Subjective Effects of Smoking Tobacco (QSU)
Description: Change from baseline Questionnaire for Urges to Smoke (post - pre).
  This is a 10-item measure where participants rate smoking-related items on a 6-point Likert scale ranging from 1 (strongly disagree) to 6 (strongly agree). Items are collapsed into two previously identified factors (Factor 1: strong desire and intention to smoke; Factor 2: anticipation of relief from withdrawal symptoms). Scores are calculated by summing the items and range from 5 to 30 with higher scores indicating greater urge to smoke.
Time Frame: Approximately 30 to 90 minutes
Population: 1 participant in the high humectant, medium sweetness arm and 1 participant in the medium humectant, medium sweetness arm declined to provide responses post-smoking.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Humectant, High Sweetness | High Humectant, Medium Sweetness | Medium Humectant, High Sweetness | Medium Humectant, Medium Sweetness
Number analyzed (Participants) | 47 | 45 | 46 | 47
score on a scale
  Desire | -7.28 (6.30) | -9.16 (6.63) | -7.22 (6.14) | -7.66 (6.49)
  Relief | -2.13 (3.84) | -2.38 (4.14) | -2.46 (4.55) | -2.23 (3.96)

15. Primary Outcome: Change in Nicotine Withdrawal Assessment (MNWS)
Description: Change from baseline using Waterpipe-modified Minnesota Withdrawal Scale (post - pre).
  The scale ranges from 0 (not at all) to 100 (extremely) with higher total numbers meaning greater withdrawal symptoms.
Time Frame: Approximately 30 to 90 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Humectant, High Sweetness | High Humectant, Medium Sweetness | Medium Humectant, High Sweetness | Medium Humectant, Medium Sweetness
Number analyzed (Participants) | 47 | 46 | 46 | 48
score on a scale
  Urges to Smoke a Waterpipe | -15.64 (26.68) | -25.15 (27.80) | -17.02 (27.51) | -20.17 (26.92)
  Irritability/Frustration/Anger | -6.94 (15.46) | -2.26 (14.56) | -2.17 (10.28) | -5.25 (17.87)
  Anxious | -5.51 (16.11) | -2.65 (10.47) | -2.85 (12.81) | -2.88 (14.83)
  Difficulty Concentrating | -5.72 (19.01) | -2.30 (10.61) | -4.46 (16.99) | -5.27 (20.12)
  Restlessness | -4.68 (18.51) | -5.63 (17.58) | -0.13 (13.45) | -2.88 (13.89)
  Hunger | 6.04 (26.84) | 6.87 (24.78) | 5.48 (20.38) | 5.31 (21.76)
  Impatient | -5.19 (16.35) | -3.13 (11.19) | -2.17 (19.07) | -1.92 (18.80)
  Craving a Waterpipe/Nicotine | -15.55 (26.68) | -19.70 (28.96) | -14.17 (30.12) | -13.13 (29.38)
  Drowsiness | -4.38 (16.61) | -5.83 (11.58) | -3.74 (16.36) | -1.17 (12.37)
  Depression/Feeling Blue | -3.15 (11.53) | -2.59 (7.74) | -3.24 (12.43) | -2.71 (10.06)
  Desire for Sweets | -6.23 (20.27) | -1.85 (17.83) | -2.15 (11.32) | -1.98 (16.84)

16. Primary Outcome: Tobacco Flavor Perception (gLMS)
Description: To determine the relative intensity of specific flavors, e.g., sweetness, the general version of the Labeled Magnitude Scale (gLMS) was used post-smoking session. The scale ranges from 0 to 100 where higher scores indicate that the perception is stronger.
Time Frame: Post Smoking Session
Population: One participant declined to provide a response during their the high humectant, high sweetness study visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Humectant, High Sweetness | High Humectant, Medium Sweetness | Medium Humectant, High Sweetness | Medium Humectant, Medium Sweetness
Number analyzed (Participants) | 46 | 46 | 46 | 48
score on a scale
  Sweetness | 10.65 (9.50) | 9.29 (10.77) | 9.83 (11.50) | 11.64 (11.72)
  Bitterness | 18.93 (16.45) | 24.65 (18.19) | 20.93 (18.10) | 26.27 (20.83)
  Smoothness | 23.20 (15.84) | 19.54 (16.36) | 20.70 (18.40) | 17.52 (11.34)
  Harshness | 15.09 (12.76) | 21.72 (20.15) | 19.74 (17.20) | 25.79 (24.77)
  Coolness | 10.41 (12.63) | 10.04 (14.47) | 8.18 (9.90) | 7.29 (9.41)

17. Primary Outcome: Tobacco Flavors Perception, Degree of Liking or Disliking (LHS)
Description: To assess the degree of liking or disliking of flavors, will use the Labeled Hedonic Scale (LHS) to collect ratio-level data on the magnitude of liking and disliking of sensation post-smoking session. Scores range from 0 to 100 with higher scores indicating greater liking.
Time Frame: Post Smoking Session
Population: One participant declined to provide a response during their the high humectant, high sweetness study visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Humectant, High Sweetness | High Humectant, Medium Sweetness | Medium Humectant, High Sweetness | Medium Humectant, Medium Sweetness
Number analyzed (Participants) | 46 | 46 | 46 | 48
score on a scale | 37.43 (12.57) | 32.15 (13.17) | 34.37 (14.49) | 30.38 (14.67)

18. Primary Outcome: Puffing Topography - Puff Volume
Description: Puff volume measured continuously during the smoking session using the research-grade waterpipe.
Time Frame: Up to 60 minutes
Measure: Mean (Standard Deviation); unit: Liters
Units Other Than Participants: Puffs
Arm/Group | High Humectant, High Sweetness | High Humectant, Medium Sweetness | Medium Humectant, High Sweetness | Medium Humectant, Medium Sweetness
Number analyzed (Participants) | 47 | 46 | 46 | 48
Number analyzed (Puffs) | 3025 | 2218 | 2650 | 2383
Liters | 0.72 (0.48) | 0.63 (0.46) | 0.74 (0.52) | 0.64 (0.47)

19. Primary Outcome: Puffing Topography - Puff Duration
Description: Puff duration measured continuously during the smoking session using the research-grade waterpipe.
Time Frame: Up to 60 minutes
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: Puffs
Arm/Group | High Humectant, High Sweetness | High Humectant, Medium Sweetness | Medium Humectant, High Sweetness | Medium Humectant, Medium Sweetness
Number analyzed (Participants) | 47 | 46 | 46 | 48
Number analyzed (Puffs) | 3025 | 2218 | 2650 | 2383
seconds | 3.43 (1.99) | 3.04 (1.78) | 3.62 (2.28) | 3.19 (1.85)

20. Primary Outcome: Puffing Topography - Flow Rate
Description: Puffing average flow rate measured continuously during the smoking session using the research-grade waterpipe.
Time Frame: Up to 60 minutes
Measure: Mean (Standard Deviation); unit: Liters / Minute
Units Other Than Participants: Puffs
Arm/Group | High Humectant, High Sweetness | High Humectant, Medium Sweetness | Medium Humectant, High Sweetness | Medium Humectant, Medium Sweetness
Number analyzed (Participants) | 47 | 46 | 46 | 48
Number analyzed (Puffs) | 3025 | 2218 | 2650 | 2383
Liters / Minute | 12.11 (4.29) | 11.66 (4.50) | 11.81 (3.96) | 11.24 (3.63)

21. Primary Outcome: Puffing Topography - Peak Flow Rate
Description: Puffing peak flow rate measured continuously during the smoking session using the research-grade waterpipe.
Time Frame: Up to 60 minutes
Measure: Mean (Standard Deviation); unit: Liters / Minute
Units Other Than Participants: Puffs
Arm/Group | High Humectant, High Sweetness | High Humectant, Medium Sweetness | Medium Humectant, High Sweetness | Medium Humectant, Medium Sweetness
Number analyzed (Participants) | 47 | 46 | 46 | 48
Number analyzed (Puffs) | 3025 | 2218 | 2650 | 2383
Liters / Minute | 14.57 (5.37) | 13.93 (5.68) | 14.18 (4.92) | 13.37 (4.56)

22. Primary Outcome: Puffing Topography - Interpuff Interval
Description: Interpuff interval measured continuously during the smoking session using the research-grade waterpipe.
Time Frame: Up to 60 minutes
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: Puffs
Arm/Group | High Humectant, High Sweetness | High Humectant, Medium Sweetness | Medium Humectant, High Sweetness | Medium Humectant, Medium Sweetness
Number analyzed (Participants) | 47 | 46 | 46 | 48
Number analyzed (Puffs) | 3025 | 2218 | 2650 | 2383
seconds | 21.01 (36.65) | 27.73 (53.68) | 23.69 (44.55) | 27.90 (48.96)

ADVERSE EVENTS:
Time Frame: Approximately 1 Month
Arm/Group | High Humectant, High Sweetness | High Humectant, Medium Sweetness | Medium Humectant, High Sweetness | Medium Humectant, Medium Sweetness
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/46 | 0/46 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/46 | 0/46 | 0/48
Other Adverse Events (participants affected / at risk) | 0/47 | 0/46 | 0/46 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-05-03): https://cdn.clinicaltrials.gov/large-docs/73/NCT05453773/Prot_SAP_ICF_000.pdf